CLINICAL TRIAL: NCT04548154
Title: Proximal Resistance Training to Improve Walking Capacity and Physical Activity in People With Multiple Sclerosis: A Feasibility Study
Brief Title: Proximal Resistance Training for People With Multiple Sclerosis
Acronym: PT-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-1527; K12HD055931 (NIH)
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Hip abduction; Trunk muscles
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proximal Resistance Training (Experimental): Participants will receive 6 one-on-one supervised intervention visits and 8 telerehabilitation visits over 10 weeks. For the first 4 weeks intervention frequency will start with 1x/ week in clinic and 1x/ week via telerehabilitation, and the participant will be asked to perform exercises 2x/ week independently. For the final 6 weeks there will be 1x week supervised visits (weeks 6 and 8 in person, and weeks 5,7, 9, and 10 via telerehabilitation) and the participant will be asked to perform exercises 3x/ week independently.
  Interventions: Other: Proximal Resistance Training

INTERVENTIONS:
Other: Proximal Resistance Training — Participants will be prescribed 5 categories of resistance exercises, and each category will have a series of exercises to select from. Two will target hip abduction, two will target trunk muscles, and one will target functional resistance training for the hip and trunk during walking-related tasks such as multi-directional resisted walking. Dosing will be based on guidelines for MS. Strengthening exercises will begin with 3 sets of 12-15 reps at 15 rep-max load (RM) and progress to 3 sets of 8-10 reps at 10-12 RM. Endurance exercises requiring a static hold will progress from 3 sets of 15-20 second holds to 30-second holds. Functional resistance will be dosed to improve muscular endurance: 3 sets of 15-20 reps based on form fatigue.

SUMMARY:
The objective of this study is to pilot a 10-week resistance and functional movement intervention targeting proximal muscles in 40 people with MS. The investigators will assess implementation feasibility (recruitment, fidelity, retention, satisfaction), collect pilot data for key walking function outcomes, and examine movement-pattern and activity behavior mechanisms. Walking function will be measured by walking capacity (6-Minute Walk Test - 6MWT) and PA quantity (average steps/ day over 10 days). Movement-pattern mechanisms will be measured using 3D motion capture analysis (pelvis and trunk kinematics). Activity behavior mechanisms will be measured by patient-reported outcome questionnaires (perception of walking ability, self-efficacy, and readiness to change).

DETAILED DESCRIPTION:
The proposed study will be a prospective cohort in 40 people with MS with one baseline and one follow-up assessment after a 10-week functional resistance training intervention. The screening and outcome assessments will take place in the CU Interdisciplinary Movement Science Lab and intervention will occur in the CU Physical Therapy Program gym. Both facilities have the necessary space and equipment for outcomes assessment and intervention, respectively. The PI will perform the initial screening and deliver the intervention. In order to limit testing bias, all functional tests, patient-reported outcomes, and motion capture data collection will be performed by an experienced research assistant.

Participants will receive 14 one-on-one supervised intervention visits over 10 weeks. Intervention frequency will mimic clinical practice, starting at 2x/ week in clinic (2x/ week independently) for four weeks and tapering to 1x/ week in clinic (3x/ week independently) for the final six weeks. Participants will be prescribed 5 categories of resistance exercises, and each category will have a series of exercises to select from. Two will target hip abduction (lying down and standing), two will target trunk muscles (sidelying/ forward planks, resisted trunk rotation), and one will target functional resistance training for the hip and trunk during walking-related tasks such as multi-directional resisted walking. Dosing will be based on guidelines for MS. Strengthening exercises will begin with 3 sets of 12-15 reps at 15 rep-max load (RM) and progress to 3 sets of 8-10 reps at 10-12 RM. Endurance exercises requiring a static hold will progress from 3 sets of 15-20 second holds to 30-second holds. Functional resistance will be dosed to improve muscular endurance: 3 sets of 15-20 reps based on form fatigue. Progression will be achieved by modifying body position, and/or adding cuff weights or resistance bands. Exercises will take 30-45 minutes to complete. Upper extremity use to maintain balance will be allowed as needed.

ELIGIBILITY:
Inclusion Criteria.

* 18-64 years old
* Neurologist-confirmed diagnosis of MS
* Able to walk at least 100 meters without an assistive device
* Expanded Disability Status Scale - EDSS < 6
* Have their own tablet/phone/computer capable of video calls/Zoom meetings.

Exclusion Criteria.

* Other conditions limiting their ability to exercise or walk
* Unsafe to exercise as determined by a neurologist or physical therapist
* Currently undergoing physical therapy
* Unable to provide consent or follow simple directions
* Have an MS-related exacerbation or changes to their disease-modifying drug therapy in the month prior to enrollment
* A 25 foot walk test time of > 4.5 seconds

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walk test | Baseline, end of 10 week intervention period, 22 week follow-up.
  The 6MWT assesses walking endurance via the maximal distance an individual is able to walk in 6 minutes, reported in meters

SECONDARY OUTCOMES:
Change in average daily step count | Baseline, end of 10 week intervention period, 22 week follow-up.
  Step count will be measured by waist-mounted ActiGraph accelerometer-based activity monitors
Change in movement patterns | Baseline, end of 10 week intervention period, 22 week follow-up.
  Mechanisms of movement patterns will be measured by 3-dimensional motion capture analysis during self-selected walking speed and during a 30 second chair raise test.
Change in Multiple Sclerosis Walking Scale-12 | Baseline, end of 10 week intervention period, 22 week follow-up.
  A 12 questions assessment of self-reported walking mobility in people with multiple sclerosis. Scores range from 0 to 100 with higher scores indicating better mobility.
Change in Multiple Sclerosis Self-Efficacy Score | Baseline, end of 10 week intervention period, 22 week follow-up.
  An 18 item assessment of measures of self-efficacy in multiple sclerosis including a function component and a control component. Total score is reported on a 10-100 point scale with higher scores indicating greater certainty in ones ability to manage multiple sclerosis symptoms.
Change in Exercise Self-Efficacy Scale | Baseline, end of 10 week intervention period, 22 week follow-up.
  A 9 item questionnaire that assesses perceptions about ability to participate in at least 20 minutes of moderate physical activity 3x per week. Scores range from 0 to 90 points with higher scores indicating more confidence to exercise in different circumstances.
Change in Exercise Stages of Change category | Baseline, end of 10 week intervention period, 22 week follow-up.
  A 4 item measure to assess readiness to participate in exercise and activity. Depending on the answers to the yes/no questions, results are categorized as "pre-contemplation", "contemplation", "preparation", "action", and "maintenance".
Change in Modified Fatigue Impact Scale | Baseline, end of 10 week intervention period, 22 week follow-up.
  The standard measure of patient-reported limitations due to fatigue in people with MS. Scores range from 0 to 84 with higher scores indicating higher impact of fatigue on daily activities.

OTHER OUTCOMES:
Change in Patient-Specific Functional Scale | Baseline and end of 10 week intervention period.
  Participant identifies 3 activities that the participant is unable to do, or is difficult for the participant to do and rates them on a 10-point scale, with higher scores indicating greater ability to perform activity.
Change in hip abduction strength | Baseline, end of 10 week intervention period, 22 week follow-up.
  Hip abduction strength will be measured in kg using hand-held dynamometry.
Change in lateral trunk flexion strength | Baseline, end of 10 week intervention period, 22 week follow-up.
  Lateral trunk flexion strength will be measured in kg using hand-held dynamometry.
Change in lateral trunk flexion endurance | Baseline, end of 10 week intervention period, 22 week follow-up.
  Trunk flexion endurance as measured by a clinical trunk curl-up test which counts the number of trunk curls a participant can perform in 1 minute.
Expanding Disability Status Scale | Baseline
  Neurological exam used to assess disability in people with multiple sclerosis. Scores range from 0 to 6 with higher scores indicating more disability.
25 Foot Walk Test | Baseline and after the 10 week intervention period.
  Amount of time in seconds it takes for participant to walk 25 feet as quickly and safely as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Mark M. Manago, DPT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
We will publish the trial results data on the ClinicalTrials.gov website, on which the clinical trial will be registered. Sharing of data will include the potential of sharing raw data generated from all clinical assessments under a data-sharing agreement.
Supporting Information: ICF, CSR
Time Frame: We will publish the trial results within one year of testing the final participant.
Access Criteria: User registration will be required to access/download any data and will require agreement to conditions of use in accordance with NIH Data Sharing Policy Guidelines.

REFERENCES:
- [Derived] Manago MM, Cohen ET, Cameron MH, Christiansen CL, Bade M. Reliability, Validity, and Responsiveness of the Patient-Specific Functional Scale for Measuring Mobility-Related Goals in People With Multiple Sclerosis. J Neurol Phys Ther. 2023 Jul 1;47(3):139-145. doi: 10.1097/NPT.0000000000000439. Epub 2023 Mar 7. PMID 36897202